CLINICAL TRIAL: NCT01189929
Title: A Phase 1b Study of Gemcitabine and Demcizumab (OMP-21M18) With or Without Abraxane® as 1st-line Treatment in Subjects With Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: A Study of Gemcitabine and Demcizumab (OMP-21M18) With or Without Abraxane® as 1st-line Treatment in Subjects With Locally Advanced or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OncoMed Pharmaceuticals, Inc. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Organization: Mereo BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M18-002
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Pancreatic Cancer
Keywords: Phase 1,; dose escalation,; histologically; cytologically; confirmed; malignancy; metastatic
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — demcizumab; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine and demcizumab With or Without Abraxane® (Experimental): Gemcitabine and demcizumab With or Without Abraxane®
  Interventions: Drug: Demcizumab; Drug: Abraxane®; Drug: Gemcitabine

INTERVENTIONS:
Drug: Demcizumab — Up to 50 subjects will be enrolled at up to 8 centers in Australia, New Zealand, and Spain. Up to 28 days (4 weeks) prior to treatment you will undergo testing to determine your eligibility to take part in this study, and then if you are enrolled in the study you will receive intravenous (in the vein) infusions of the demcizumab administered once every 2 weeks, and gemcitabine and Abraxane® administered weekly for 3 weeks, out of every 4 weeks. After 9 weeks, you will undergo assessments to determine the status of your disease. If there is no evidence of progression of your disease or if your tumor is smaller, you will continue to receive one additional infusion of demcizumab, and you will continue to receive infusions of gemcitabine and Abraxane® once weekly for 3 consecutive weeks out of every 4 weeks until it has been shown that your cancer has progressed. You will undergo assessments every 8 weeks thereafter to determine the status of your disease.
  Other Names: OMP-21M18
Drug: Abraxane® — Abraxane® which will be administered by IV infusion at a dose of 125 mg/m2 over 30 minutes once a week for 3 weeks in a row, followed by a week of rest.
Drug: Gemcitabine — Gemcitabine will be administered intravenously over 30 minutes initially at a dose of 1000 mg/m2 once a week for 3 weeks in a row, followed by a week of rest. If you develop side effects during this time period, your physician may decide to hold or reduce the dose of gemcitabine.

SUMMARY:
The purpose of this study is to test the safety and determine the optimal dose of a new experimental drug, demcizumab (OMP-21M18), when given in combination with gemcitabine with or without (+/-) Abraxane®. Historically, single agent gemcitabine has been the standard treatment for pancreatic cancer. However, recent data suggests that gemcitabine plus Abraxane® may be superior to gemcitabine alone, thus this combination is emerging as the new standard therapy for pancreatic cancer. However, Abraxane® has not been approved for the treatment of pancreatic cancer at this time. Demcizumab is a humanized monoclonal antibody and was developed to target cancer stem cells. This study is sponsored by OncoMed Pharmaceuticals, which is referred to as OncoMed or the Sponsor in this consent form. The study is designed to test the safety of demcizumab at different dose levels when given with gemcitabine +/- Abraxane® and the effects, both good and bad, that it has on participants. Demcizumab may block the growth of cancer stem cells, the remaining tumor cells, and it may also prevent the growth of new blood vessels that tumors need to grow and spread. Although demcizumab has been administered with gemcitabine to cancer patients, it has not been given in combination with gemcitabine and Abraxane®; thus, it is not known if it will provide any benefit to participants and may cause harmful side effects.

DETAILED DESCRIPTION:
Current cancer therapies often produce an initial reduction in tumour size but may not have long term benefits. One possible explanation for this is the presence cancer cell known as a cancer stem cells. Cancer stem cells represent a small part of the tumour but are believed to be responsible for much of the growth and spread of the cancer. They may also be more resistant to traditional therapy, such as chemotherapy and radiation therapy.

The purpose of this study is to test the safety and determine the optimal dose of a new experimental drug, demcizumab, when given in combination with gemcitabine, a drug that is a standard treatment for advanced pancreatic cancer that has not been treated previously with chemotherapy. Demcizumab is a humanized monoclonal antibody (a protein made in the laboratory) and was developed to target cancer stem cells. The way the body handles demcizumab will also be investigated.

Up to 50 subjects will be enrolled at up to 8 centers in Australia, New Zealand, and Spain. Up to 28 days (4 weeks) prior to treatment you will undergo testing to determine your eligibility to take part in this study, and then if you are enrolled in the study you will receive intravenous (in the vein) infusions of the demcizumab administered once every 2 weeks, and gemcitabine and Abraxane® administered weekly for 3 weeks, out of every 4 weeks. After 9 weeks, you will undergo assessments to determine the status of your disease. If there is no evidence of progression of your disease or if your tumor is smaller, you will continue to receive one additional infusion of demcizumab, and you will continue to receive infusions of gemcitabine and Abraxane® once weekly for 3 consecutive weeks out of every 4 weeks until it has been shown that your cancer has progressed. You will undergo assessments every 8 weeks thereafter to determine the status of your disease. If there is no evidence of progression of your disease or if your tumor is smaller, you will continue to receive one additional infusion of demcizumab, and you will continue to receive infusions of gemcitabine and Abraxane® once weekly for 3 consecutive weeks out of every 4 weeks until it has been shown that your cancer has progressed. You will undergo assessments every 8 weeks thereafter to determine the status of your disease.

In addition to routine testing of blood and urine (for complete blood counts with differential and platelets, coagulation studies to determine how quickly your blood is clotting , serum chemistries, B-type natriuretic peptide [BNP] and Troponin I which indicates how well your heart if working, and urinalysis), special tests will be performed during the study at specific time points.

In addition, you will have and ECG and Doppler echocardiogram performed during screening, then every 28 days on study and at treatment termination. Your Doppler echocardiograms may be sent to a Cardiologist at another hospital who may perform a central read on some of the Doppler echocardiograms in this study. Finally, you will have a head CT or MRI at baseline and CT scans and/or other radiographs performed every 56 days to assess the status of your tumor.

The study includes an optional part which will investigate how variations in people's genetic makeup affect their response to medications. This involves the collection of one blood sample just before participants receive their first dose of study treatment. DNA will be extracted from the blood sample for testing.

ELIGIBILITY:
Inclusion criteria

1. Subjects must have histologically or cytologically confirmed locally advanced or metastatic pancreatic cancer. In addition, subjects must have a tumor that is at least 1 cm in a single dimension and is radiographically apparent on Computed Topography (CT) or Magnetic Resonance Imaging (MRI). Prior chemotherapy or radiotherapy is not allowed.
2. Age >21 years
3. Eastern Cooperative Oncology Group (ECOG) performance status <2 (see Appendix B)
4. Life expectancy of more than 3 months
5. Subjects must have normal organ and marrow function as defined below:

   * Leukocytes >3.5 x 109/L
   * Absolute neutrophil count >1.25 x 109/L
   * Hemoglobin >100 g/L
   * Platelets >125 X 109/L
   * Total bilirubin <2 X institutional upper limit of normal (ULN)
   * Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) <5 X institutional ULN
   * Alkaline phosphatase <5 X institutional ULN
   * International normalized ratio (INR) and activated partial thromboplastin time (aPTT) within institutional ULN
   * Creatinine <1.5 X institutional ULN OR
   * Calculated creatinine clearance >60 mL/min using the Cockcroft and Gault formula as follows:

   Creatinine clearance (mL/min) = (140 - age) x ideal body weight [kg] 0.814 x serum creatinine [µmol/L] For women, multiply the value from the equation above by 0.85. Where age is in years, weight is in kg, and serum creatinine is in µmol/L
6. Women of childbearing potential must have had a prior hysterectomy or have a negative serum pregnancy test and be using adequate contraception prior to study entry and must agree to use adequate contraception from study entry through at least 6 months after discontinuation of study drug. Men must also agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and from study entry through at least 6 months after discontinuation of study drug. Should a woman enrolled in the study or a female partner of a man enrolled in the study become pregnant or suspect she is pregnant while participating in this study or within 6 months after discontinuation of study drug, the Investigator should be informed immediately.
7. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria

Subjects who meet any of the following criteria will not be eligible for participation in the study:

1. Subjects receiving any other investigational agents or anti-cancer therapy.
2. Subjects with brain metastases (subjects must have a CT scan or MRI of the head within 28 days prior to enrollment to rule out brain metastases), uncontrolled seizure disorder, or active neurologic disease
3. History of a significant allergic reaction attributed to humanized or human monoclonal antibody therapy
4. Significant intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
5. Pregnant women or nursing women
6. Subjects with known HIV infection
7. Known bleeding disorder or coagulopathy
8. Subjects receiving heparin, warfarin, or other similar anticoagulants. Note: Subjects may be receiving low-dose aspirin and/or non-steroidal anti-inflammatory agents.
9. Subjects with known clinically significant gastrointestinal disease including, but not limited to, inflammatory bowel disease
10. New York Heart Association Classification II, III, or IV
11. Subjects with a blood pressure (BP) of >140/90 mmHg. Subjects taking antihypertensive medications must be taking ≤2 medications to obtain this level of BP control.
12. Subjects with tumors that are currently involving the lumen of the gastrointestinal tract
13. Subjects with current evidence of cardiac ischemia or heart failure within the last 6 months, subjects who are receiving any medications for cardiac ischemia, subjects with a B-type natriuretic peptide (BNP) value of >100 pg/mL, subjects with a LVEF of <50%, subjects with pulmonary hypertension defined as a peak tricuspid velocity >3.4 m/s on doppler echocardiogram or subjects that have received a total cumulative dose of ≥400 mg/m2 doxorubicin
14. Subjects with electrocardiogram (ECG) evidence of ischemia or ≥ Grade 2 ventricular arrhythmia, subjects who have a history of acute myocardial infarction within 6 months, or subjects with unstable angina

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of demcizumab (OMP-21M18) when combined with gemcitabine +/- Abraxane® | Until disease progression

SECONDARY OUTCOMES:
To determine the safety of gemcitabine +/- Abraxane® plus demcizumab (OMP-21M18) | Until disease progression
To determine the rate of immunogenicity of gemcitabine +/- Abraxane® plus demcizumab (OMP-21M18) | Until disease progression
To determine the preliminary efficacy of gemcitabine +/- Abraxane® plus demcizumab (OMP-21M18) | Until disease progression
To determine population pharmacokinetics of demcizumab (OMP-21M18) | Until disease progression
To determine the exploratory biomarker changes of gemcitabine plus demcizumab (OMP-21M18) | Until disease progression

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Box Hill Hospital, Box Hill, Victoria
  - The Austin Hospital, Heidelberg, Victoria
- New Zealand (2):
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton
- START Madrid, Madrid, Spain